CLINICAL TRIAL: NCT03232983
Title: Effect of Injection Site on the Relative and Absolute Bioavailability of Single Dose of LY900014 in Healthy Subjects
Brief Title: A Study of LY900014 Formulation at Different Injection Sites in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 16639; I8B-MC-ITRT (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-07-26; First posted 2017-07-28 (Actual); Results first posted 2020-04-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2017-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- LY900014 (SC Abdomen) (Experimental): Single dose of 15-U of LY900014 administered subcutaneously (SC) into the abdomen in one period
  Interventions: Drug: LY900014 (SC)
- LY900014 (SC Thigh) (Experimental): Single dose of 15-U of LY900014 administered SC into the thigh in one period
  Interventions: Drug: LY900014 (SC)
- LY900014 (SC Arm) (Experimental): Single dose of 15-U of LY900014 administered SC into the arm (deltoid) in one period
  Interventions: Drug: LY900014 (SC)
- LY900014 (IV) (Active Comparator): Single dose of 15-U of LY900014 administered intravenously (IV) in one period
  Interventions: Drug: LY900014 (IV)

INTERVENTIONS:
Drug: LY900014 (SC) — Administered SC
  Other Names: Ultra-Rapid Lispro
  Arms: LY900014 (SC Abdomen); LY900014 (SC Arm); LY900014 (SC Thigh)
Drug: LY900014 (IV) — Administered IV
  Other Names: Ultra-Rapid Lispro
  Arms: LY900014 (IV)

SUMMARY:
This study evaluates a new formulation of insulin lispro, LY900014, a drug that lowers blood sugar. It is administered by injection into the vein and under the skin of the abdomen, thigh and arm.

The study will be conducted in healthy people to investigate the effect of different injection sites on the amount of insulin lispro in the bloodstream.

Side effects and tolerability will be documented. The study will last for about 10 weeks for each participant, including screening and follow up. Screening is required within 28 days prior to entering the study.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy male or a female (not pregnant and agreeable to take birth control measures until study completion)
* Have a body mass index (BMI) of 18 to 30 kilogram per square meter (kg/m²)
* Have normal blood pressure, pulse rate, electrocardiogram (ECG), blood and urine laboratory test results that are acceptable for the study
* Are nonsmokers, have not smoked for at least 6 months prior to entering the study

Exclusion Criteria:

* Are currently participating in or completed a clinical trial within the last 30 days or any other type of medical research judged to be incompatible with this study
* Have previously participated or withdrawn from this study
* Had blood loss of more than 450 milliliters (mL) within the last 3 months

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2017-11-09 (Actual); Study Completion 2017-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Singapore, Singapore

REFERENCES:
- [Derived] Leohr JK, Dellva MA, LaBell E, Coutant DE, Linnebjerg H. Evaluation of the Pharmacokinetic Profile of Ultra Rapid Lispro Administered Subcutaneously at Different Injection Sites. Clin Ther. 2022 Jun;44(6):836-847. doi: 10.1016/j.clinthera.2022.04.001. Epub 2022 May 13. PMID 35577602

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is an open-label, randomized, crossover, up to 10-hour euglycemic clamp study in which participants were randomized into one of four treatment sequences. Participants received single doses of 15 units of LY900014 on 4 occasions (treatment Periods 1 through 4) with a wash-out period of at least 3 days between study drug administration.
Groups:
- LY900014 Treatment Sequence 1: Abdomen,Thigh, Deltoid(Arm), IV: Single dose of 15-U of LY900014 administered subcutaneously (SC) into the abdomen in Period 1, Thigh in Period 2, Deltoid (Arm) in Period 3, and single 15-U intravenous (IV) bolus injection in Period 4.
- LY900014 Treatment Sequence 2: Deltoid, Abdomen, IV, Thigh: Single dose of 15-U of LY900014 administered SC into the: Deltoid in Period 1, Abdomen in Period 2, single 15-U IV bolus injection in Period 3, and single 15-U SC administration into the Thigh in Period 4.
- LY900014 Treatment Sequence 3: IV, Deltoid, Thigh, Abdomen: Single 15-U IV bolus injection of LY900014 administered in Period 1, single 15-U dose administered SC in the Deltoid in Period 2, Thigh in Period 3, and Abdomen in Period 4.
- LY900014 Treatment Sequence 4: Thigh, IV, Abdomen, Deltoid: Single dose of 15-U of LY900014 administered SC in Thigh in Period 1, single 15-U IV bolus injection in Period 2, single dose of 15-U administered SC in the Abdomen in Period 3, and Deltoid in Period 4.
Period: Period 1
Arm/Group | LY900014 Treatment Sequence 1: Abdomen,Thigh, Deltoid(Arm), IV | LY900014 Treatment Sequence 2: Deltoid, Abdomen, IV, Thigh | LY900014 Treatment Sequence 3: IV, Deltoid, Thigh, Abdomen | LY900014 Treatment Sequence 4: Thigh, IV, Abdomen, Deltoid
Started | 7 | 7 | 7 | 7
Received at Least One Dose of Study Drug | 7 | 7 | 7 | 7
Completed | 7 | 7 | 6 | 7
Not Completed | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Period: Washout Period 1
Arm/Group | LY900014 Treatment Sequence 1: Abdomen,Thigh, Deltoid(Arm), IV | LY900014 Treatment Sequence 2: Deltoid, Abdomen, IV, Thigh | LY900014 Treatment Sequence 3: IV, Deltoid, Thigh, Abdomen | LY900014 Treatment Sequence 4: Thigh, IV, Abdomen, Deltoid
Started | 7 | 7 | 6 | 7
Completed | 7 | 7 | 6 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | LY900014 Treatment Sequence 1: Abdomen,Thigh, Deltoid(Arm), IV | LY900014 Treatment Sequence 2: Deltoid, Abdomen, IV, Thigh | LY900014 Treatment Sequence 3: IV, Deltoid, Thigh, Abdomen | LY900014 Treatment Sequence 4: Thigh, IV, Abdomen, Deltoid
Started | 7 | 7 | 6 | 7
Completed | 7 | 7 | 6 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 2
Arm/Group | LY900014 Treatment Sequence 1: Abdomen,Thigh, Deltoid(Arm), IV | LY900014 Treatment Sequence 2: Deltoid, Abdomen, IV, Thigh | LY900014 Treatment Sequence 3: IV, Deltoid, Thigh, Abdomen | LY900014 Treatment Sequence 4: Thigh, IV, Abdomen, Deltoid
Started | 7 | 7 | 6 | 7
Completed | 7 | 7 | 5 | 6
Not Completed | 0 | 0 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Period: Period 3
Arm/Group | LY900014 Treatment Sequence 1: Abdomen,Thigh, Deltoid(Arm), IV | LY900014 Treatment Sequence 2: Deltoid, Abdomen, IV, Thigh | LY900014 Treatment Sequence 3: IV, Deltoid, Thigh, Abdomen | LY900014 Treatment Sequence 4: Thigh, IV, Abdomen, Deltoid
Started | 7 | 7 | 5 | 6
Completed | 7 | 7 | 5 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 3
Arm/Group | LY900014 Treatment Sequence 1: Abdomen,Thigh, Deltoid(Arm), IV | LY900014 Treatment Sequence 2: Deltoid, Abdomen, IV, Thigh | LY900014 Treatment Sequence 3: IV, Deltoid, Thigh, Abdomen | LY900014 Treatment Sequence 4: Thigh, IV, Abdomen, Deltoid
Started | 7 | 7 | 5 | 6
Completed | 7 | 7 | 5 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | LY900014 Treatment Sequence 1: Abdomen,Thigh, Deltoid(Arm), IV | LY900014 Treatment Sequence 2: Deltoid, Abdomen, IV, Thigh | LY900014 Treatment Sequence 3: IV, Deltoid, Thigh, Abdomen | LY900014 Treatment Sequence 4: Thigh, IV, Abdomen, Deltoid
Started | 7 | 7 | 5 | 6
Completed | 6 | 7 | 5 | 6
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants.
Groups:
- Overall: Single 15-U dose of LY900014 administered in treatment Period 1- 4, as SC injection into the abdomen, the thigh, the deltoid or an IV bolus injection, per randomized treatment sequence.
Arm/Group | Overall
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 28
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 28
Weight [Geometric Mean (Standard Deviation); unit: kilograms (kg)] | 70.11 (10.48)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Insulin Lispro Area Under the Concentration Versus Time Curve (AUC) Following LY900014 Administration
Description: Pharmacokinetics(PK): Insulin lispro AUC from time zero to 10 hours post dose [AUC(0-10h)].
Time Frame: Day 1: Pre-dose, 2.5, 5, 10, 15, 20, 25, 30, 40, 60, 70, 90, 120, 150, 180, 210, 240, 300, 360, 420, 480, 540, and 600 minutes post-dose
Population: All participants who have received at least one dose of study drug and have measurable insulin lispro concentrations and evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomole * hour/Liter (pmol * hr/L)
Groups:
- LY900014 (SC Abdomen): Single 15-U dose of LY900014 administered subcutaneously (SC) into the abdomen in one period.
- LY900014 (SC Deltoid): Single 15-U dose of LY900014 administered SC into the deltoid in one period.
- LY900014 (IV): Single 15-U injection IV bolus of LY900014 administered in one period.
- LY900014 (SC Thigh): Single 15-U dose of LY900014 administered SC into the thigh in one period.
Arm/Group | LY900014 (SC Abdomen) | LY900014 (SC Deltoid) | LY900014 (IV) | LY900014 (SC Thigh)
Number analyzed (Participants) | 25 | 26 | 27 | 26
picomole * hour/Liter (pmol * hr/L) | 1760 (20) | 1800 (16) | 2770 (22) | 1750 (19)
Statistical Analysis 1: Comparison: LY900014 (SC Abdomen) vs LY900014 (SC Deltoid); Geometric Least Squares Means (LSMeans) were controlled for injection site, study period, and sequence as fixed effects, and subject within sequence as a random effect; Test type: Superiority; Mixed Models Analysis; Ratio of Geometric Least Squares Means = 1.03, 90% CI 2-sided [0.992 to 1.07]
Statistical Analysis 2: Comparison: LY900014 (SC Abdomen) vs LY900014 (SC Thigh); Geometric LSMeans were controlled for injection site, study period, and sequence as fixed effects, and subject within sequence as a random effect; Test type: Superiority; Mixed Models Analysis; Ratio of Geometric Least Squares Means = 1.00, 90% CI 2-sided [0.962 to 1.04]

2. Secondary Outcome: Total Amount of Glucose Infused (Gtot) Over Duration of the Clamp Procedure
Description: Glucodynamics: Gtot is the total glucose infusion over the clamp duration (10 hours) and is used to measure the study drug action over time as measured by the euglycemic clamp procedure. During the euglycemic clamp procedure, blood glucose concentrations are held constant after the administration of LY900014 by adjusting the exogenous glucose infusion rate.
Time Frame: Every 10 minutes for 30 minutes predose, every 2.5 minutes for 30 minutes, then every 5 minutes for 120 minutes, then every 10 minutes for 120 to 480 minutes and every 10 minutes for 480 to 600 minutes post-dose
Population: All participants who have received at least one dose of study drug administered and have completed at least one clamp procedure. The IV treatment arm was needed only for PK as it served as the reference to determine the absolute bioavailability.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: milligram per kilogram (mg/kg)
Groups:
- LY900014 (SC Deltoid): Single 15-U dose of LY900014 administered SC into the arm in one period.
Arm/Group | LY900014 (SC Abdomen) | LY900014 (SC Deltoid) | LY900014 (SC Thigh)
Number analyzed (Participants) | 25 | 26 | 26
milligram per kilogram (mg/kg) | 1490 (45) | 1630 (50) | 1730 (38)
Statistical Analysis 1: Comparison: LY900014 (SC Abdomen) vs LY900014 (SC Deltoid); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Mixed Models Analysis; Ratio of Geometric LSMeans = 1.09, 90% CI 2-sided [1.00 to 1.20]
Statistical Analysis 2: Comparison: LY900014 (SC Abdomen) vs LY900014 (SC Thigh); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Mixed Models Analysis; Ratio of Geometric LSMeans = 1.14, 90% CI 2-sided [1.04 to 1.25]

ADVERSE EVENTS:
Time Frame: Baseline to end of study (up to 49 days)
Description: All participants who received at least one dose of study drug.
Groups:
- 15-U LY900014 Abdomen: Single dose of 15-U of LY900014 administered subcutaneously (SC) into the abdomen.
- 15-U LY900014 Thigh: Single dose of 15-U of LY900014 administered SC into the Thigh.
- 15-U LY900014 Deltoid: Single dose of 15-U of LY900014 administered SC into the Deltoid.
- 15-U LY900014 IV: Single 15-U LY900014 administered IV bolus injection.
Arm/Group | 15-U LY900014 Abdomen | 15-U LY900014 Thigh | 15-U LY900014 Deltoid | 15-U LY900014 IV
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/26 | 0/26 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/26 | 0/26 | 0/28
Other Adverse Events (participants affected / at risk) | 6/25 | 7/26 | 11/26 | 4/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15-U LY900014 Abdomen (N=25) | 15-U LY900014 Thigh (N=26) | 15-U LY900014 Deltoid (N=26) | 15-U LY900014 IV (N=28)
Application site erythema (General disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (2)
Catheter site bruise (General disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (2)
Catheter site erythema (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Catheter site pain (General disorders) | 1 (2) | 1 (1) | 1 (1) | 3 (4)
Catheter site swelling (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Infusion site erythema (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Infusion site pain (General disorders) | 3 (4) | 0 (0) | 1 (1) | 1 (1)
Infusion site swelling (General disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Injection site pain (General disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Vessel puncture site bruise (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/83/NCT03232983/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-04): https://cdn.clinicaltrials.gov/large-docs/83/NCT03232983/SAP_001.pdf